CLINICAL TRIAL: NCT00664495
Title: Reduction of Abdominal Obesity and Insulin Resistance in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Queen's University
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Ross 1999
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Obesity
Keywords: Obesity, exercise, diet, insulin resistance
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance | interventions — Diet, Reducing; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- C (No Intervention): Control
- DWL (Active Comparator): Diet Weight Loss
  Interventions: Behavioral: Diet Weight Loss
- EWL (Active Comparator): Exercise Weight Loss
  Interventions: Behavioral: Exercise Weight Loss
- EWS (Active Comparator): Exercise Without Weight Loss
  Interventions: Behavioral: Exercise Without Weight Loss

INTERVENTIONS:
Behavioral: Diet Weight Loss
  Arms: DWL
Behavioral: Exercise Weight Loss
  Arms: EWL
Behavioral: Exercise Without Weight Loss
  Arms: EWS

SUMMARY:
The purpose of the study was to assess the effects of equivalent diet- or exercise-induced weight loss and related insulin resistance in abdominally obese women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women

Exclusion Criteria:

* Smokers and diabetics

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 1999-04; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Abdominal Obesity | 4 months
Insulin Resistance | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Result] Ross R, Janssen I, Dawson J, Kungl AM, Kuk JL, Wong SL, Nguyen-Duy TB, Lee S, Kilpatrick K, Hudson R. Exercise-induced reduction in obesity and insulin resistance in women: a randomized controlled trial. Obes Res. 2004 May;12(5):789-98. doi: 10.1038/oby.2004.95. PMID 15166299